CLINICAL TRIAL: NCT06106776
Title: PROSPECTIVE OBSERVATIONAL STUDY FOR THE ASSESSMENT OF CARDIAC DYSFUNCTION INDUCED BY CHIMERIC ANTIGEN RECEPTOR T (CAR-T) CELL THERAPY
Brief Title: CAR-T Cell Induced Cardiac Dysfunction: A Prospective Study
Acronym: CARdio-Tox
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6000
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Receptors, Chimeric Antigen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chimeric Antigen Receptor — This study will evaluate the incidence of cardiac dysfunction at 7 days and 1 month after chimeric antigen receptor-T cell infusion (tisagenlecleucel, axicabtagene ciloleucel e brexucabtagene autoleucel).

SUMMARY:
In this observational, prospective study, patients affected by B-cell Lymphoma and candidate to chimeric antigen receptor-T (CAR-T) cell infusion will be evaluated at three timepoints to establish the rate of cardiac dysfunction, defined according to 2022 European Society of Cardiology Cardio-Oncology guidelines. Echocardiography, physical examination and cardiac/inflammatory biomarkers will be performed prior to CAR-T cell infusion and followed at 7 days and 1 month.

DETAILED DESCRIPTION:
Patients will perform clinical evaluation, transthoracic echocardiogram with speckle tracking analysis and blood samples (including cardiac biomarkers of damage and fibrosis) prior to CART infusion, after 7 days and 1 month following CART infusion. Rate of Cytokine Release Syndrome and use of interleukin-6 inhibitors will be also registered.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old;
* Patients affected by relapsed and/or refractory diffuse large B-cell lymphoma, follicular lymphoma, primary mediastinal B-cell lymphoma, mantle cell lymphoma or B-cell lymphoblastic leukemia, candidate treatment with chimeric antigen receptor-T cell therapy at the Hematology division of Policlinico Universitario Agostino Gemelli, Rome;
* Patients with left ventricular ejection fraction >50%.

Exclusion Criteria:

* Age<18 years old;
* Patients who denied to participate to the study;
* Patients with left ventricular ejection fraction<50%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by relapsed and/or refractory diffuse large B-cell lymphoma, follicular lymphoma, primary mediastinal B-cell lymphoma, mantle cell lymphoma or B-cell lymphoblastic leukemia, scheduled to receive treatment with chimeric antigen receptor-T cell therapy at the Hematology division of Policlinico Universitario Agostino Gemelli, Rome will be firstly evaluated. If they exclusion criteria are not present, the will be included in the study protocol and evaluated by the Cardio-Oncology outpatient service.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2023-11-02 (Estimated); Primary Completion 2024-11-02 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Cancer Therapy Related Cardiac Dysfunction | 30 days
  Cancer Therapy Related Cardiac Dysfunction will be defined according to 2022 European Society of Cardiology guidelines, as symptomatic or asymptomatic and mild, moderate or severe.

SECONDARY OUTCOMES:
Correlation with Inflammatory Biomarkers | 30 days
  Modifications of echocardiographic metrics will be related to inflammatory biomarkers (interleukin2 soluble receptor, interleukin 6, fibrinogen, C-reactive protein) changes.
Correlation with Cytokine Release Syndrome Occurrence | 30 days
  Incidence of cardiotoxicity will be related to occurrence and severity of Cytokine Release Syndrome